CLINICAL TRIAL: NCT03048422
Title: Phase III Study of the Virologic Efficacy and Safety of Dolutegravir-Containing Versus Efavirenz-Containing Antiretroviral Therapy Regimens in HIV-1-Infected Pregnant Women and Their Infants
Brief Title: Evaluating the Efficacy and Safety of Dolutegravir-Containing Versus Efavirenz-Containing Antiretroviral Therapy Regimens in HIV-1-Infected Pregnant Women and Their Infants
Acronym: VESTED
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMPAACT 2010; 30129 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2017-02-07; First posted 2017-02-09 (Estimated); Results first posted 2021-11-10 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — dolutegravir; emtricitabine tenofovir alafenamide; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Efavirenz, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm 1: Maternal DTG+FTC/TAF (Experimental): Mothers randomized to receive dolutegravir (DTG) plus emtricitabine/tenofovir alafenamide (FTC/TAF) during pregnancy, through delivery, and for 50 weeks postpartum.
  Interventions: Drug: Dolutegravir; Drug: Emtricitabine/tenofovir alafenamide
- Arm 2: Maternal DTG+FTC/TDF (Experimental): Mothers randomized to receive DTG plus emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) during pregnancy, through delivery, and for 50 weeks postpartum.
  Interventions: Drug: Dolutegravir; Drug: Emtricitabine/tenofovir disoproxil fumarate
- Arm 3: Maternal EFV/FTC/TDF (Active Comparator): Mothers randomized to receive efavirenz/emtricitabine/tenofovir disoproxil fumarate (EFV/FTC/TDF) during pregnancy, through delivery, and for 50 weeks postpartum.
  Interventions: Drug: Efavirenz/emtricitabine/tenofovir disoproxil fumarate
- Arm 1 Infants (No Intervention): Infants born to women in Arm 1. Infants did not directly receive study intervention, but may have been exposed to the randomized treatment through placental or breastmilk transfer.
- Arm 2 Infants (No Intervention): Infants born to women in Arm 2. Infants did not directly receive study intervention, but may have been exposed to the randomized treatment through placental or breastmilk transfer.
- Arm 3 Infants (No Intervention): Infants born to women in Arm 3. Infants did not directly receive study intervention, but may have been exposed to the randomized treatment through placental or breastmilk transfer.

INTERVENTIONS:
Drug: Dolutegravir — One 50 mg DTG tablet was administered orally once daily
  Other Names: DTG
  Arms: Arm 1: Maternal DTG+FTC/TAF; Arm 2: Maternal DTG+FTC/TDF
Drug: Emtricitabine/tenofovir alafenamide — One fixed-dose combination tablet (FTC 200 mg/TAF 25 mg) was administered orally once daily
  Other Names: FTC/TAF
  Arms: Arm 1: Maternal DTG+FTC/TAF
Drug: Emtricitabine/tenofovir disoproxil fumarate — One fixed-dose combination tablet (FTC 200 mg/TDF 300 mg) was administered orally once daily
  Other Names: FTC/TDF
  Arms: Arm 2: Maternal DTG+FTC/TDF
Drug: Efavirenz/emtricitabine/tenofovir disoproxil fumarate — One fixed-dose combination tablet (EFV 600 mg/FTC 200 mg/TDF 300 mg) was administered orally once daily
  Other Names: EFV/FTC/TDF
  Arms: Arm 3: Maternal EFV/FTC/TDF

SUMMARY:
The purpose of this study was to compare the virologic efficacy and safety of three antiretroviral (ARV) regimens, dolutegravir plus emtricitabine/tenofovir alafenamide, dolutegravir plus emtricitabine/tenofovir disoproxil fumarate, and efavirenz/emtricitabine/tenofovir disoproxil fumarate in pregnant women living with HIV-1 and to compare the safety of these regimens for their infants.

DETAILED DESCRIPTION:
This study compared the virologic efficacy and safety of three ARV regimens in pregnant women living with HIV: dolutegravir (DTG) plus emtricitabine/tenofovir alafenamide (FTC/TAF), DTG plus emtricitabine/tenofovir disoproxil fumarate (FTC/TDF), and efavirenz/emtricitabine/tenofovir disoproxil fumarate (EFV/FTC/TDF). The study also compared the safety of these regimens for their infants.

At study entry, mothers were randomly assigned to either receive DTG plus FTC/TAF (Arm 1), DTG plus FTC/TDF (Arm 2), or EFV/FTC/TDF (Arm 3) during pregnancy, through delivery, and for 50 weeks postpartum.

Mothers completed study visits at study entry and every four weeks during pregnancy. Study visits for mothers and their infants occurred at delivery and at 6, 14, 26, 38, and 50 weeks postpartum. Visits for mothers and infants included physical examinations and blood collection. Select study visits also included breast milk collection from mothers who breastfed, hair and urine collection, ultrasound scans, pregnancy testing, contraception counseling, and, for a subset of participants, dual energy x-ray absorptiometry (DXA) scans for mothers and their infants.

For pregnancy outcome measures, mothers and infants were evaluated together as mother-infant pairs, with any outcome between the two counting as an event (for example, if an infant was born small for gestational age, this would be a pregnancy outcome event for the mother-infant pair). For all other outcome measures, women and infants were evaluated separately.

ELIGIBILITY:
Inclusion Criteria:

* Mother is able to provide written informed consent for her and her infant's participation in this study
* Mother has confirmed HIV-1 infection based on documented testing of two samples collected at different time points:

  * Sample #1 may be tested using any of the following:
  * Two rapid antibody tests from different manufacturers or based on different principles and epitopes
  * One enzyme immunoassay (EIA) OR Western blot OR immunofluorescence assay OR chemiluminescence assay
  * One HIV DNA polymerase chain reaction (PCR)
  * One quantitative HIV RNA PCR (above the limit of detection of the assay)
  * One qualitative HIV RNA PCR
  * One total HIV nucleic acid test
  * Sample #2 may be tested using any of the following:
  * One rapid antibody test. If this option is used in combination with two rapid tests for Sample #1, at least one of the three rapid tests must be FDA-approved and the third rapid test must be from a third manufacturer or based on a third principle or epitope.
  * One EIA OR Western blot OR immunofluorescence assay OR chemiluminescence assay
  * One HIV DNA PCR
  * One quantitative HIV RNA PCR (above the limit of detection of the assay)
  * One qualitative HIV RNA PCR
  * One total HIV nucleic acid test.
  * See the protocol for more information on this inclusion criterion.
* At screening, mother is ART-naive, defined as having not received prior antiretroviral therapy other than ARVs received during prior pregnancies or prior periods of breastfeeding (i.e., receipt of any single, dual, or triple ARV regimen during prior time-limited periods of pregnancy and breastfeeding is permitted). Receipt of up to 14 days of ARVs during the current pregnancy is permitted prior to study entry so that initiation of ARVs during the current pregnancy is not delayed during the study screening period. Note: Non-study ART may be initiated in the current pregnancy prior to initiation of the study screening process. For eligible participants, enrollment must occur within 14 days of non-study ART initiation. Note: Receipt of ARVs during a prior pregnancy or prior period of breastfeeding must have concluded at least six months prior to study entry. Receipt of TDF or FTC/TDF for pre-exposure prophylaxis at any time in the past is not exclusionary (even if received within six months prior to study entry).
* At screening, mother has the following laboratory test results (based on testing of samples collected within 14 days prior to study entry):

  * Grade 1 or lower (less than 2.5 times upper limit of normal [ULN]) alanine aminotransferase (ALT) and aspartate aminotransferase (AST)
  * Grade 2 or lower (less than or equal to 1.8 times ULN) creatinine
  * Grade 2 or lower (greater than or equal to 60 mL/min) estimated creatinine clearance (CrCl; Cockcroft-Gault formula). See the protocol for guidance on severity grading. Laboratory tests may be repeated during the study screening period, with the latest result used for eligibility determination.
* At screening and at study entry, no evidence of multiple gestation or fetal anomalies, as assessed by best available method
* At study entry, gestational age of 14-28 weeks, defined as greater than 13 weeks plus six days and less than 28 completed weeks gestation, estimated by best available method. Note: For this inclusion criterion and the previous inclusion criterion, fetal ultrasound is preferred but not required for purposes of eligibility determination. If ultrasound cannot be performed during the study screening period prior to study entry, it must be performed within 14 days after study entry. As further explained in the protocol, enrolled participants will not be withdrawn from the study based on ultrasound findings obtained after study entry.
* At study entry, mother expects to remain in the geographic area of the study site during pregnancy and for 50 weeks postpartum [Eligibility criteria added per Letter of Amendment 1 to V2; July 2018]:
* At study entry, mother reports that she does not wish to become pregnant again for at least 50 weeks after her current pregnancy and that she is willing to use effective contraception during this period. Effective contraception may include surgical sterilization (i.e., hysterectomy, bilateral oophorectomy, tubal ligation, or salpingectomy) or any of the following methods:

  * Contraceptive intrauterine device (IUD) or intrauterine system (IUS)
  * Subdermal contraceptive implant
  * Progestogen injections
  * Progestogen only oral contraceptive pills
  * Combined estrogen and progestogen oral contraceptive pills
  * Percutaneous contraceptive patches
  * Contraceptive vaginal rings
  * Note: IUDs, IUSs, implants, and injections are strongly recommended due to their lower failure rates with typical use. Male or female condom use is recommended with all contraceptive methods for dual protection against pregnancy and to avoid transmission of HIV and other sexually transmitted infections.

Exclusion Criteria:

* Mother is currently incarcerated or involuntarily confined in a medical facility
* Mother is currently receiving:

  * A psychoactive medication for treatment of a psychiatric illness
  * Treatment for active tuberculosis
  * Treatment for active hepatitis C infection
* Mother is expected to require treatment with interferon and/or ribavirin for hepatitis C infection during the study follow-up period
* Mother has a history of any of the following, as determined by the site investigator or designee based on maternal report and available medical records:

  * Hypersensitivity or clinically significant adverse reaction to any of the ARVs included in the three study drug regimens (ever)
  * Antiretroviral drug resistance mutations that would impact selection of ART regimen (ever)
  * Clinically significant heart disease and/or known prolonged corrected QT (QTc) interval (ever)
  * Suicidal ideation or attempt (ever)
  * HIV-2 infection (ever)
  * Zika virus infection, diagnosed or suspected, during the current pregnancy
  * Receipt of any antiretroviral medication within six months prior to study entry, with two exceptions: receipt of any duration of TDF or FTC/TDF for pre-exposure prophylaxis or receipt of up to 14 days of ARVs during the current pregnancy
  * Receipt of any prohibited medication within 14 days prior to study entry (see the protocol for more information)
  * Clinically significant acute illness requiring systemic treatment and/or hospitalization (i.e., major medical condition that is likely to lead to hospitalization and/or to an adverse pregnancy outcome) within 14 days prior to study entry
  * Unstable liver disease (defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice) or known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones) within 14 days prior to study entry
  * Note: Testing to rule out HIV-2 infection is not required.
* Mother or fetus has any other condition that, in the opinion of the site investigator or designee, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 643 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2020-10-03 (Actual); Study Completion 2020-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shahin Lockman, MD, MSc, Study Chair — Harvard T.H. Chan School of Public Health and Brigham and Women's Hospital; Lameck Chinula, MBBS, MMED, FCOG, Study Chair — Kamuzu Central Hospital in Lilongwe, Malawi
Locations (21):
- United States (2):
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Pediatric Perinatal HIV Clinical Trials Unit CRS, Miami, Florida
- Botswana (2):
  - Gaborone CRS, Gaborone, South-East District
  - Molepolole CRS, Gaborone
- Brazil (4):
  - SOM Federal University Minas Gerais Brazil NICHD CRS, Belo Horizonte, Minas Gerais
  - Hospital Federal dos Servidores do Estado NICHD CRS, Rio de Janeiro
  - Instituto de Puericultura e Pediatria Martagao Gesteira - UFRJ NICHD CRS, Rio de Janeiro
  - Hosp. Geral De Nova Igaucu Brazil NICHD CRS, Rio de Janeiro
- Byramjee Jeejeebhoy Medical College (BJMC) CRS, Pune, Maharashtra, India
- South Africa (4):
  - Soweto IMPAACT CRS, Johannesburg, Gauteng
  - Wits RHI Shandukani Research Centre CRS, Johannesburg, Gauteng
  - Umlazi CRS, Durban, KwaZulu-Natal
  - Famcru Crs, Tygerberg, Western Cape
- Kilimanjaro Christian Medical Centre (KCMC), Moshi, Tanzania
- Thailand (3):
  - Siriraj Hospital ,Mahidol University NICHD CRS, Bangkok, Bangkoknoi
  - Chiangrai Prachanukroh Hospital NICHD CRS, Chiang Mai
  - Chiang Mai University HIV Treatment (CMU HIV Treatment) CRS, Chiang Mai
- Baylor-Uganda CRS, Kampala, Uganda
- Zimbabwe (3):
  - Seke North CRS, Chitungwiza
  - St Mary's CRS, Chitungwiza
  - Harare Family Care CRS, Harare

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the International Maternal Pediatric Adolescent AIDS Clinical Trial (IMPAACT) Network by NIH
Access Criteria: * With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the IMPAACT Network.
  * For what types of analyses? To achieve aims in the proposal approved by the IMPAACT Network.
  * By what mechanism will data be made available? Researchers may submit a request for access to data using the IMPAACT "Data Request" form at: https://www.impaactnetwork.org/studies/submit-research-proposal. Researchers of approved proposals will need to sign an IMPAACT Data Use Agreement before receiving the data.
URL: https://www.impaactnetwork.org/studies/submit-research-proposal

REFERENCES:
- [Result] Lockman S, Brummel SS, Ziemba L, Stranix-Chibanda L, McCarthy K, Coletti A, Jean-Philippe P, Johnston B, Krotje C, Fairlie L, Hoffman RM, Sax PE, Moyo S, Chakhtoura N, Stringer JS, Masheto G, Korutaro V, Cassim H, Mmbaga BT, Joao E, Hanley S, Purdue L, Holmes LB, Momper JD, Shapiro RL, Thoofer NK, Rooney JF, Frenkel LM, Amico KR, Chinula L, Currier J; IMPAACT 2010/VESTED Study Team and Investigators. Efficacy and safety of dolutegravir with emtricitabine and tenofovir alafenamide fumarate or tenofovir disoproxil fumarate, and efavirenz, emtricitabine, and tenofovir disoproxil fumarate HIV antiretroviral therapy regimens started in pregnancy (IMPAACT 2010/VESTED): a multicentre, open-label, randomised, controlled, phase 3 trial. Lancet. 2021 Apr 3;397(10281):1276-1292. doi: 10.1016/S0140-6736(21)00314-7. PMID 33812487
- [Derived] Masheto G, Brummel SS, Ziemba L, Shepherd J, Mbengeranwa T, Igawa L, Coletti A, Mukura D, Rossouw L, Theron G, Krotje C, Jean-Philippe P, Chakhtoura N, Cassim H, Mathiba SR, Maena J, Murtaugh W, Fairlie L, Currier J, Hoffman R, Chinula L, Sax PE, Stranix-Chibanda L, Lockman S; IMPAACT 2010/VESTED Study Team and Investigators. Markers of Maternal Bone and Renal Toxicity Through 50 Weeks Postpartum: IMPAACT 2010 (VESTED) Trial. J Acquir Immune Defic Syndr. 2024 Oct 1;97(2):172-179. doi: 10.1097/QAI.0000000000003478. PMID 39250651
- [Derived] Eke AC, Brummel SS, Aliyu MH, Stranix-Chibanda L, Eleje GU, Ezebialu IU, Korutaro V, Wabwire D, Matubu A, Mbengeranwa T, Chakhtoura N, Chinula L, McCarthy K, Knowles K, Krotje C, Linton MF, Dooley KE, Sax PE, Brown T, Lockman S; IMPAACT 2010/VESTED Study Team. Lipid and Glucose Profiles in Pregnant Women With HIV on Tenofovir-based Antiretroviral Therapy. Clin Infect Dis. 2025 Mar 17;80(3):594-601. doi: 10.1093/cid/ciae441. PMID 39219495
- [Derived] Jacobson DL, Crider KS, DeMarrais P, Brummel S, Zhang M, Pfeiffer CM, Moore CA, McCarthy K, Johnston B, Mohammed T, Vhembo T, Kabugho E, Muzorah GA, Cassim H, Fairlie L, Machado ES, Ngocho JS, Shapiro RL, Serghides L, Chakhtoura N, Chinula L, Lockman S. Dolutegravir- Versus Efavirenz-Based Treatment in Pregnancy: Impact on Red Blood Cell Folate Concentrations in Pregnant Women and Their Infants. J Infect Dis. 2024 Nov 15;230(5):1224-1234. doi: 10.1093/infdis/jiae308. PMID 38877762
- [Derived] Chinula L, Ziemba L, Brummel S, McCarthy K, Coletti A, Krotje C, Johnston B, Knowles K, Moyo S, Stranix-Chibanda L, Hoffman R, Sax PE, Stringer J, Chakhtoura N, Jean-Philippe P, Korutaro V, Cassim H, Fairlie L, Masheto G, Boyce C, Frenkel LM, Amico KR, Purdue L, Shapiro R, Mmbaga BT, Patel F, van Wyk J, Rooney JF, Currier JS, Lockman S; IMPAACT 2010/VESTED Study Team and Investigators. Efficacy and safety of three antiretroviral therapy regimens started in pregnancy up to 50 weeks post partum: a multicentre, open-label, randomised, controlled, phase 3 trial. Lancet HIV. 2023 Jun;10(6):e363-e374. doi: 10.1016/S2352-3018(23)00061-9. Epub 2023 May 8. PMID 37167996
- See also: Study website — http://impaactnetwork.org/studies/impaact2010
- See also: The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017, was used — http://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables
- See also: Intergrowth 21st Standards, including reference for infants small for gestational age — http://intergrowth21.tghn.org/standards-tools/
- See also: FDA Snapshot algorithm — http://www.fda.gov/files/drugs/published/Human-Immunodeficiency-Virus-1-Infection--Developing-Antiretroviral-Drugs-for-Treatment.pdf
- See also: Definition for major congenital anomalies — http://pubmed.ncbi.nlm.nih.gov/21800414/
- See also: Schwartz formula for calculating infant creatinine clearance — http://www-users.med.cornell.edu/~spon/picu/calc/crclschw.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Maternal DTG+FTC/TAF: Mothers randomized to receive DTG+FTC/TAF
- Arm 2: Maternal DTG+FTC/TDF: Mothers randomized to receive DTG+FTC/TDF
- Arm 3: Maternal EFV/FTC/TDF: Mothers randomized to receive EFV/FTC/TDF
Period: Overall Study
Arm/Group | Arm 1: Maternal DTG+FTC/TAF | Arm 2: Maternal DTG+FTC/TDF | Arm 3: Maternal EFV/FTC/TDF
Started | 217 | 215 | 211
Completed | 200 | 205 | 202
Not Completed | 17 | 10 | 9
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 5 | 0 | 1
Not completed — Withdrawal by Subject | 5 | 7 | 4
Not completed — Moved | 3 | 2 | 2
Not completed — Noncompliant with Study Requirements | 2 | 1 | 2
Not completed — Not Able to Get to Clinic | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Enrolled women.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Maternal DTG+FTC/TAF | Arm 2: Maternal DTG+FTC/TDF | Arm 3: Maternal EFV/FTC/TDF | Total
Number analyzed (Participants) | 217 | 215 | 211 | 643
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.5 (6.2) | 27.0 (5.8) | 27.7 (5.9) | 27.4 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 217 | 215 | 211 | 643
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 21 | 18 | 60
  Not Hispanic or Latino | 194 | 192 | 190 | 576
  Unknown or Not Reported | 2 | 2 | 3 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 195 | 196 | 194 | 585
  Race: Asian | 7 | 5 | 6 | 18
  Race: Other | 10 | 6 | 4 | 20
  Race: White | 5 | 7 | 7 | 19
  Race: Unknown | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 2 | 0 | 4
  Botswana | 16 | 18 | 17 | 51
  Tanzania | 15 | 13 | 15 | 43
  Brazil | 21 | 19 | 17 | 57
  South Africa | 37 | 37 | 37 | 111
  Uganda | 37 | 37 | 36 | 110
  Zimbabwe | 82 | 84 | 83 | 249
  Thailand | 5 | 4 | 6 | 15
  India | 2 | 1 | 0 | 3
Gestational Age [Mean (Standard Deviation); unit: weeks] | 21.6 (4.2) | 21.4 (4.2) | 21.8 (4.2) | 21.6 (4.2)
Gestational Age Stratification Group [Count of Participants; unit: Participants]
  14-18 Weeks | 58 | 64 | 59 | 181
  19-23 Weeks | 93 | 83 | 77 | 253
  24-28 Weeks | 66 | 68 | 75 | 209
Plasma HIV-1 RNA Viral Load [Mean (Standard Deviation); unit: copies/mL] — Population: Plasma HIV RNA viral load among participants who had baseline viral load data available.
  copies/mL
    number analyzed (Participants) | 216 | 215 | 209 | 640
    (all) | 14,558.2 (45,813.9) | 18,420.3 (97,896.4) | 13,381.2 (42,042.5) | 15,471.2 (67,050.5)
Plasma HIV-1 RNA Viral Load <200 copies/mL [Count of Participants; unit: Participants] — Population: Participants with plasma HIV-1 RNA viral load data available at baseline
  Participants
    number analyzed (Participants) | 216 | 215 | 209 | 640
    (all) | 62 | 66 | 53 | 181
Weight [Mean (Standard Deviation); unit: kg] | 67.7 (15.1) | 66.3 (16.8) | 64.5 (13.3) | 66.2 (15.2)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Mothers With HIV-1 RNA Viral Load Less Than 200 Copies/mL at Delivery
Description: Percentage of mothers with plasma HIV-1 RNA viral load less than 200 copies/mL at delivery determined using real-time test results obtained at site laboratories. This outcome was evaluated in the non-inferiority (primary outcome) and superiority (secondary outcome) analyses. The intention-to-treat analysis included all randomized women who had viral load data available. The per-protocol analysis excluded women who modified randomized treatment (stopped, paused, switched, added any treatment) before viral load evaluation at delivery, with the exception of women who modified randomized treatment for use of a concomitant medication.
Time Frame: Delivery
Population: Women who had plasma HIV-1 RNA viral load data available at delivery
Measure: Number; unit: Percentage of participants
Groups:
- Arms 1 and 2: Maternal DTG+FTC/TAF and DTG+FTC/TDF: Combined group of mothers randomized to receive dolutegravir DTG+FTC/TAF or DTG+FTC/TDF
Arm/Group | Arms 1 and 2: Maternal DTG+FTC/TAF and DTG+FTC/TDF | Arm 3: Maternal EFV/FTC/TDF
Number analyzed (Participants) | 405 | 200
Percentage of participants
  Intention-to-Treat Analysis | 97.5 | 91.0
  Per-Protocol Analysis | 97.5 | 91.4
Statistical Analysis 1: Comparison: Arms 1 and 2: Maternal DTG+FTC/TAF and DTG+FTC/TDF vs Arm 3: Maternal EFV/FTC/TDF; Difference in proportions for intention-to-treat analysis; Test type: Non-Inferiority — Equivalence margin was a 10% difference between groups; Risk Difference (RD) = 6.5, 95% CI 2-sided [2.0 to 10.7]
Statistical Analysis 2: Comparison: Arms 1 and 2: Maternal DTG+FTC/TAF and DTG+FTC/TDF vs Arm 3: Maternal EFV/FTC/TDF; Difference in proportions for per-protocol analysis; Test type: Non-Inferiority — Equivalence margin was a 10% difference between groups; Risk Difference (RD) = 6.0, 95% CI 2-sided [1.6 to 10.3]
Statistical Analysis 3: Comparison: Arms 1 and 2: Maternal DTG+FTC/TAF and DTG+FTC/TDF vs Arm 3: Maternal EFV/FTC/TDF; Difference in proportions for superiority and intention-to-treat analysis; Test type: Superiority; p = 0.005, Wald test of two proportions; Risk Difference (RD) = 6.5, 95% CI 2-sided [2.0 to 10.7]

2. Primary Outcome: Percentage of Mother-infant Pairs With an Adverse Pregnancy Outcome
Description: Percentage of mother-infant pairs with an adverse pregnancy outcome. Adverse pregnancy outcome includes spontaneous abortion (<20 weeks gestation), stillbirth (≥20 weeks gestation), preterm delivery (<37 completed weeks), or small for gestational age (<10th percentile by INTERGROWTH 21st Standards)
Time Frame: Delivery
Population: Mother-infant pairs with pregnancy outcome evaluated on study.
Measure: Number; unit: percentage of mother-infant pairs
Arm/Group | Arm 1: Maternal DTG+FTC/TAF | Arm 2: Maternal DTG+FTC/TDF | Arm 3: Maternal EFV/FTC/TDF
Number analyzed (Participants) | 216 | 213 | 211
percentage of mother-infant pairs | 24.1 | 32.9 | 32.7
Statistical Analysis 1: Comparison: Arm 1: Maternal DTG+FTC/TAF vs Arm 2: Maternal DTG+FTC/TDF; Null hypothesis of no difference between groups (DTG+FTC/TAF - DTG+FTC/TDF); Test type: Superiority; p = 0.043, Wald test of two proportions; Risk Difference (RD) = -8.8, 95% CI 2-sided [-17.3 to -0.3]
Statistical Analysis 2: Comparison: Arm 2: Maternal DTG+FTC/TDF vs Arm 3: Maternal EFV/FTC/TDF; Null hypothesis of no difference between groups (DTG+FTC/TDF - EFV/FTC/TDF); Test type: Superiority; p = 0.97, Wald test of two proportions; Risk Difference (RD) = 0.2, 95% CI 2-sided [-8.8 to 9.1]
Statistical Analysis 3: Comparison: Arm 1: Maternal DTG+FTC/TAF vs Arm 3: Maternal EFV/FTC/TDF; Null hypothesis of no difference between groups (DTG+FTC/TAF - EFV/FTC/TDF); Test type: Superiority; p = 0.047, Wald test of two proportions; Risk Difference (RD) = -8.6, 95% CI 2-sided [-17.1 to -0.1]

3. Primary Outcome: Cumulative Probability of Women Experiencing Grade 3 or Higher Adverse Event
Description: The Kaplan-Meier estimate of the cumulative probability of women experiencing grade 3 or higher adverse events, including events resulting in death due to any cause.
  Time to first maternal grade 3 or higher adverse event was defined as the first grade 3 or higher adverse event that occurred after randomization and before 74 weeks of follow-up. The timeframe of 74 weeks was determined by adding up 56 weeks of postpartum follow-up to the mean duration of antepartum follow-up, which was 18 weeks.
Time Frame: From randomization up to 74 weeks
Population: Enrolled women.
Measure: Number; unit: Cumulative probability per 100 persons
Arm/Group | Arm 1: Maternal DTG+FTC/TAF | Arm 2: Maternal DTG+FTC/TDF | Arm 3: Maternal EFV/FTC/TDF
Number analyzed (Participants) | 217 | 215 | 211
Cumulative probability per 100 persons | 25.1 | 30.8 | 27.9
Statistical Analysis 1: Comparison: Arm 1: Maternal DTG+FTC/TAF vs Arm 2: Maternal DTG+FTC/TDF; The Kaplan-Meier method was used to estimate survival probabilities. Survival probabilities were compared based on a Z-test using Greenwoods estimate of the standard error. The null hypothesis was no difference between arms (DTG+FTC/TAF - DTG+FTC/TDF); Test type: Superiority; p = 0.098, Z-test; Risk Difference (RD) = -5.6, 95% CI 2-sided [-14.2 to 2.9]
Statistical Analysis 2: Comparison: Arm 2: Maternal DTG+FTC/TDF vs Arm 3: Maternal EFV/FTC/TDF; The Kaplan-Meier method was used to estimate survival probabilities. Survival probabilities were compared based on a Z-test using Greenwoods estimate of the standard error. The null hypothesis was no difference between arms (DTG+FTC/TDF-EFV/FTC/TDF); Test type: Superiority; p = 0.26, Z-test; Risk Difference (RD) = 2.6, 95% CI 2-sided [-5.9 to 11.7]
Statistical Analysis 3: Comparison: Arm 1: Maternal DTG+FTC/TAF vs Arm 3: Maternal EFV/FTC/TDF; The Kaplan-Meier method was used to estimate survival probabilities. Survival probabilities were compared based on a Z-test using Greenwoods estimate of the standard error. The null hypothesis was no difference between arms (DTG+FTC/TAF-EFV/FTC/TDF); Test type: Superiority; p = 0.26, Z-test; Risk Difference (RD) = -2.8, 95% CI 2-sided [-11.3 to 5.8]

4. Primary Outcome: Cumulative Probability of Infants Experiencing Grade 3 or Higher Adverse Event
Description: The Kaplan-Meier estimate of the cumulative probability of infants experiencing grade 3 or higher adverse events, including events resulting in death due to any cause.
Time Frame: From birth through Week 50 postpartum
Population: Live born infants
Measure: Number; unit: Cumulative probability per 100 persons
Groups:
- Arm 1 Infants: Infants born to women who were randomized to receive DTG+FTC/TAF during pregnancy and postpartum
- Arm 2 Infants: Infants born to women who were randomized to receive DTG+FTC/TDF during pregnancy and postpartum
- Arm 3 Infants: Infants born to women who were randomized to receive EFV/FTC/TDF during pregnancy and postpartum
Arm/Group | Arm 1 Infants | Arm 2 Infants | Arm 3 Infants
Number analyzed (Participants) | 208 | 202 | 207
Cumulative probability per 100 persons | 25.3 | 28.6 | 30.9
Statistical Analysis 1: Comparison: Arm 1 Infants vs Arm 2 Infants; The Kaplan-Meier method was used to estimate survival probabilities. Comparisons of survival probabilities was based on a Z-test using Greenwoods estimate of the standard error. The null hypothesis was no difference between arms, with estimated difference of DTG+FTC/TAF - DTG+FTC/TDF; Test type: Superiority; p = 0.25, Z-test; Risk Difference (RD) = -3.2, 95% CI 2-sided [-12.8 to 6.3]
Statistical Analysis 2: Comparison: Arm 2 Infants vs Arm 3 Infants; The Kaplan-Meier method was used to estimate survival probabilities. Comparisons of survival probabilities was based on a Z-test using Greenwoods estimate of the standard error. The null hypothesis was no difference between arms, with estimate of risk difference DTG+FTC/TDF-EFV/FTC/TDF; Test type: Superiority; p = 0.32, Z-test; Risk Difference (RD) = -2.3, 95% CI 2-sided [-12.1 to 7.5]
Statistical Analysis 3: Comparison: Arm 1 Infants vs Arm 3 Infants; The Kaplan-Meier method was used to estimate survival probabilities. Comparisons of survival probabilities was based on a Z-test using Greenwoods estimate of the standard error. The null hypothesis was no difference between arms, with estimate of risk difference DTG+FTC/TAF-EFV/FTC/TDF; Test type: Superiority; p = 0.11, Z-test; Risk Difference (RD) = -5.5, 95% CI 2-sided [-14.3 to 3.2]

5. Secondary Outcome: Percentage of Mothers With HIV-1 RNA Less Than 50 Copies/mL at Delivery Measured at Central Laboratory
Description: Percentage of mothers with HIV-1 RNA less than 50 copies/mL at delivery using batched test results obtained from central laboratory
Time Frame: Delivery
Population: Women with viral load data available from central laboratory
Measure: Number; unit: percentage of participants
Arm/Group | Arms 1 and 2: Maternal DTG+FTC/TAF and DTG+FTC/TDF | Arm 3: Maternal EFV/FTC/TDF
Number analyzed (Participants) | 377 | 184
percentage of participants | 94.4 | 78.8
Statistical Analysis 1: Comparison: Arms 1 and 2: Maternal DTG+FTC/TAF and DTG+FTC/TDF vs Arm 3: Maternal EFV/FTC/TDF; Difference in proportions between arms for intention-to-treat analysis with null hypothesis of no difference (DTG groups - EFV/FTC/TDF); Test type: Superiority; p < 0.0001, Wald test of two proportions; Risk Difference (RD) = 15.6, 95% CI 2-sided [9.3 to 22.0]

6. Secondary Outcome: Percentage of Mothers With HIV-1 RNA Less Than 200 Copies/mL at 50 Weeks Postpartum
Description: Percentage of mothers with HIV-1 RNA less than 200 copies/mL at 50 weeks postpartum using real-time test results obtained from site laboratories
Time Frame: 50 weeks postpartum
Population: Women with viral load data available.
Measure: Number; unit: percentage of participants
Arm/Group | Arms 1 and 2: Maternal DTG+FTC/TAF and DTG+FTC/TDF | Arm 3: Maternal EFV/FTC/TDF
Number analyzed (Participants) | 380 | 193
percentage of participants | 96.3 | 96.4
Statistical Analysis 1: Comparison: Arms 1 and 2: Maternal DTG+FTC/TAF and DTG+FTC/TDF vs Arm 3: Maternal EFV/FTC/TDF; Difference in proportions for intention-to-treat analysis with null hypothesis of no difference between arms (DTG arms - EFV/FTC/TDF); Test type: Superiority; p = 0.97, Wald test of two proportions; Risk Difference (RD) = -0.1, 95% CI 2-sided [-3.3 to 3.2]

7. Secondary Outcome: Time to First HIV-1 RNA Less Than 200 Copies/mL Through Delivery
Description: Time to first viral HIV-1 RNA less than 200 copies/mL through delivery, determined using real-time results obtained from site laboratories
Time Frame: Randomization to delivery
Population: Women with viral load data available.
Measure: Mean (Standard Error); unit: weeks
Arm/Group | Arms 1 and 2: Maternal DTG+FTC/TAF and DTG+FTC/TDF | Arm 3: Maternal EFV/FTC/TDF
Number analyzed (Participants) | 430 | 210
weeks | 4.26 (0.09) | 6.49 (0.31)
Statistical Analysis 1: Comparison: Arms 1 and 2: Maternal DTG+FTC/TAF and DTG+FTC/TDF vs Arm 3: Maternal EFV/FTC/TDF; Test type: Superiority; p < 0.001, Kaplan-Meier; Hazard Ratio (HR) = 2.4, 95% CI 2-sided [1.9 to 3.1]

8. Secondary Outcome: Percentage of Mothers With Virologic Success of HIV-1 RNA Less Than 200 Copies/mL at Delivery Based on FDA Snapshot Algorithm
Description: Percentage of mothers with virologic success of HIV-1 RNA less than 200 copies/mL at delivery based on FDA snapshot algorithm using real-time test results obtained from site laboratories
Time Frame: Delivery
Population: Enrolled women
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Maternal DTG+FTC/TAF | Arm 2: Maternal DTG+FTC/TDF | Arm 3: Maternal EFV/FTC/TDF
Number analyzed (Participants) | 217 | 215 | 211
percentage of participants | 88.9 | 92.6 | 81.0
Statistical Analysis 1: Comparison: Arm 1: Maternal DTG+FTC/TAF vs Arm 2: Maternal DTG+FTC/TDF; Difference between arms with null hypothesis of no difference (DTG+FTC/TAF - DTG+FTC/TDF); Test type: Superiority; p = 0.19, Wald test of two proportions; Risk Difference (RD) = 3.6, 95% CI 2-sided [-1.8 to 9.1]
Statistical Analysis 2: Comparison: Arm 2: Maternal DTG+FTC/TDF vs Arm 3: Maternal EFV/FTC/TDF; Difference between arms with null hypothesis of no difference (DTG+FTC/TDF - EFV/FTC/TDF); Test type: Superiority; p < 0.001, Wald test of two proportions; Risk Difference (RD) = -11.5, 95% CI 2-sided [-17.9 to -5.2]
Statistical Analysis 3: Comparison: Arm 1: Maternal DTG+FTC/TAF vs Arm 3: Maternal EFV/FTC/TDF; Difference between arms with null hypothesis of no difference (DTG+FTC/TAF - EFV/FTC/TDF); Test type: Superiority; p = 0.022, Wald test of two proportions; Risk Difference (RD) = -7.9, 95% CI 2-sided [-14.6 to -1.2]

9. Secondary Outcome: Percentage of Mothers With Virologic Success of HIV-1 RNA Less Than 200 Copies/mL at 50 Weeks Postpartum Based on FDA Snapshot Algorithm
Description: Percentage of mothers with virologic success of HIV-1 RNA less than 200 copies/mL at 50 weeks postpartum based on FDA snapshot algorithm using real-time test results obtained from site laboratories
Time Frame: 50 weeks postpartum
Population: Enrolled women
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Maternal DTG+FTC/TAF | Arm 2: Maternal DTG+FTC/TDF | Arm 3: Maternal EFV/FTC/TDF
Number analyzed (Participants) | 217 | 215 | 211
percentage of participants | 75.6 | 77.7 | 76.3
Statistical Analysis 1: Comparison: Arm 1: Maternal DTG+FTC/TAF vs Arm 2: Maternal DTG+FTC/TDF; Difference between arms with null hypothesis of no difference (DTG+FTC/TAF - DTG+FTC/TDF); Test type: Superiority; p = 0.61, Wald test of two proportions; Risk Difference (RD) = 2.1, 95% CI 2-sided [-5.9 to 10.1]
Statistical Analysis 2: Comparison: Arm 2: Maternal DTG+FTC/TDF vs Arm 3: Maternal EFV/FTC/TDF; Difference between arms with null hypothesis of no difference (DTG+FTC/TDF - EFV/FTC/TDF); Test type: Superiority; p = 0.74, Wald test of two proportions; Risk Difference (RD) = -1.4, 95% CI 2-sided [-9.4 to 6.6]
Statistical Analysis 3: Comparison: Arm 1: Maternal DTG+FTC/TAF vs Arm 3: Maternal EFV/FTC/TDF; Difference between arms with null hypothesis of no difference (DTG+FTC/TAF - EFV/FTC/TDF); Test type: Superiority; p = 0.86, Wald test of two proportions; Risk Difference (RD) = 0.7, 95% CI 2-sided [-7.4 to 8.8]

10. Secondary Outcome: Percentage of Mother-Infant Pairs With an Adverse Pregnancy Outcome
Description: Percentage of mother-infant pairs with an adverse pregnancy outcome. Adverse pregnancy outcome includes spontaneous abortion (<20 weeks gestation), stillbirth (≥20 weeks gestation), preterm delivery (<37 completed weeks), or small for gestational age (<10th percentile per INTERGROWTH 21st Standards)
Time Frame: Delivery
Population: Mother-infant pairs with pregnancy outcome evaluated on study
Measure: Number; unit: percentage of mother-infant pairs
Arm/Group | Arms 1 and 2: Maternal DTG+FTC/TAF and DTG+FTC/TDF | Arm 3: Maternal EFV/FTC/TDF
Number analyzed (Participants) | 429 | 211
percentage of mother-infant pairs | 28.4 | 32.7
Statistical Analysis 1: Comparison: Arms 1 and 2: Maternal DTG+FTC/TAF and DTG+FTC/TDF vs Arm 3: Maternal EFV/FTC/TDF; Null hypothesis of no difference between groups (DTG groups - EFV/FTC/TDF); Test type: Superiority; p = 0.27, Wald test of two proportions; Risk Difference (RD) = 4.3, 95% CI 2-sided [-3.4 to 11.9]

11. Secondary Outcome: Cumulative Probability of Women Experiencing Grade 3 or Higher Adverse Event
Description: as for outcome 3
Time Frame: From randomization up to 74 weeks
Population: Enrolled women.
Measure: Number; unit: Cumulative probability per 100 persons
Arm/Group | Arms 1 and 2: Maternal DTG+FTC/TAF and DTG+FTC/TDF | Arm 3: Maternal EFV/FTC/TDF
Number analyzed (Participants) | 432 | 211
Cumulative probability per 100 persons | 27.9 | 27.9
Statistical Analysis 1: Comparison: Arms 1 and 2: Maternal DTG+FTC/TAF and DTG+FTC/TDF vs Arm 3: Maternal EFV/FTC/TDF; The Kaplan-Meier method was used to estimate survival probabilities. Comparisons of survival probabilities was based on a Z-test using Greenwoods estimate of the standard error. The null hypothesis was no difference between arms, with estimate of risk difference combined DTG arms-EFV/FTC/TDF; Test type: Superiority; p = 0.49, Z-test; Risk Difference (RD) = -0.1, 95% CI 2-sided [-7.6 to 7.5]

12. Secondary Outcome: Cumulative Probability of Infants Experiencing Grade 3 or Higher Adverse Event
Description: as for outcome 4
Time Frame: Birth through Week 50 postpartum
Population: Live born infants
Measure: Number; unit: Cumulative probability per 100 persons
Groups:
- Arms 1 and 2 Infants: Combined group of infants born to women who were randomized to receive DTG+FTC/TAF or DTG+FTC/TDF during pregnancy and postpartum
Arm/Group | Arms 1 and 2 Infants | Arm 3 Infants
Number analyzed (Participants) | 410 | 207
Cumulative probability per 100 persons | 26.8 | 30.9
Statistical Analysis 1: Comparison: Arms 1 and 2 Infants vs Arm 3 Infants; The Kaplan-Meier method was used to estimate survival probabilities. Comparisons of survival probabilities was based on a Z-test using Greenwoods estimate of the standard error. The null hypothesis was no difference between arms, with estimated difference of combined DTG arms - EFV/FTC/TDF; Test type: Superiority; p = 0.15, Z-test; Risk Difference (RD) = 4.1, 95% CI 2-sided [-3.8 to 12.0]

13. Secondary Outcome: Percentage of Mother-infant Pairs With an Adverse Pregnancy Outcome or Major Congenital Anomaly
Description: Percentage of mother-infant pairs with an adverse pregnancy outcome or major congenital anomaly. Adverse pregnancy outcomes include spontaneous abortions (<20 weeks gestation), stillbirths (≥20 weeks gestation), preterm deliveries (<37 weeks gestation), and infants small for gestational age (<10th percentile per INTERGROWTH 21st Standards). Major congenital anomaly was defined consistent with the definition of malformation provided by Holmes and Westgate (i.e., a structural abnormality with surgical, medical, or cosmetic importance) and evaluated by an internal study team blinded to treatment arm.
Time Frame: Delivery through 50 weeks postpartum
Population: Mother-infant pairs with pregnancy outcome evaluated on study.
Measure: Number; unit: percentage of mother-infant pairs
Arm/Group | Arm 1: Maternal DTG+FTC/TAF | Arm 2: Maternal DTG+FTC/TDF | Arm 3: Maternal EFV/FTC/TDF
Number analyzed (Participants) | 216 | 213 | 211
percentage of mother-infant pairs | 24.1 | 32.9 | 33.2
Statistical Analysis 1: Comparison: Arm 1: Maternal DTG+FTC/TAF vs Arm 2: Maternal DTG+FTC/TDF; Null hypothesis of no difference between groups (DTG+FTC/TAF - DTG+FTC/TDF); Test type: Superiority; p = 0.043, Wald test of two proportions; Risk Difference (RD) = -8.8, 95% CI 2-sided [-17.3 to -0.3]
Statistical Analysis 2: Comparison: Arm 2: Maternal DTG+FTC/TDF vs Arm 3: Maternal EFV/FTC/TDF; Null hypothesis of no difference between groups (DTG+FTC/TDF - EFV/FTC/TDF); Test type: Superiority; p = 0.95, Wald test of two proportions; Risk Difference (RD) = -0.3, 95% CI 2-sided [-9.3 to 8.6]
Statistical Analysis 3: Comparison: Arm 1: Maternal DTG+FTC/TAF vs Arm 3: Maternal EFV/FTC/TDF; Null hypothesis of no difference between groups (DTG+FTC/TAF - EFV/FTC/TDF); Test type: Superiority; p = 0.037, Wald test of two proportions; Risk Difference (RD) = -9.1, 95% CI 2-sided [-17.6 to -0.6]

14. Secondary Outcome: Count of Mother-infant Pairs in the Classified Ranked Composite Safety Outcome
Description: Infant and pregnancy outcomes were classified on a scale of 1 to 10, with mother-infant pairs categorized by the worst outcome they experienced (worst category being 1 and best being 10): 1) Infant death; 2) Spontaneous abortion (<20 weeks gestation) or stillbirth (≥20 weeks gestation); 3) Infant HIV infection; 4) Extremely and very early preterm (<32 completed weeks); 5) Major congenital anomaly; 6) Preterm delivery (<37 completed weeks); 7) Small for gestational age (<10th percentile); 8) Infant hospitalization; 9) Infant grade 3 or 4 adverse event; 10) None of the above. If a mother-infant pair experienced more than one safety outcome, only the worst was reported.
Time Frame: Birth through 50 weeks postpartum
Population: Mother-infant pairs with pregnancy outcome evaluated on study.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Maternal DTG+FTC/TAF | Arm 2: Maternal DTG+FTC/TDF | Arm 3: Maternal EFV/FTC/TDF
Number analyzed (Participants) | 216 | 213 | 211
Participants
  Infant Death | 2 | 4 | 14
  Spontaneous abortion or stillbirth | 8 | 11 | 4
  HIV-1 Infection | 2 | 0 | 1
  Extremely and Very Preterm Delivery | 1 | 1 | 2
  Major Congenital Anomaly | 2 | 0 | 1
  Preterm Delivery | 10 | 17 | 18
  Small for Gestational Age | 29 | 38 | 36
  Infant Hospitalization | 18 | 14 | 19
  Infant Grade 3 or 4 Adverse Event | 7 | 8 | 6
  None | 137 | 120 | 110
Statistical Analysis 1: Comparison: Arm 1: Maternal DTG+FTC/TAF vs Arm 2: Maternal DTG+FTC/TDF; Null hypothesis of odds ratio equal to 1, with odds of experiencing a worse outcome equal between groups (DTG+FTC/TAF - DTG+FTC/TDF); Test type: Superiority; p = 0.095, Regression, Ordinal; Odds Ratio (OR) = 0.73, 95% CI 2-sided [0.50 to 1.06]
Statistical Analysis 2: Comparison: Arm 2: Maternal DTG+FTC/TDF vs Arm 3: Maternal EFV/FTC/TDF; Null hypothesis of odds ratio equal to 1, with odds of experiencing a worse outcome equal between groups (DTG+FTC/TDF - EFV/FTC/TDF); Test type: Superiority; p = 0.30, Regression, Ordinal; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.58 to 1.19]
Statistical Analysis 3: Comparison: Arm 1: Maternal DTG+FTC/TAF vs Arm 3: Maternal EFV/FTC/TDF; Null hypothesis of odds ratio equal to 1, with odds of experiencing a worse outcome equal between groups (DTG+FTC/TAF - EFV/FTC/TDF); Test type: Superiority; p = 0.008, Regression, Ordinal; Odds Ratio (OR) = 0.60, 95% CI 2-sided [0.42 to 0.88]

15. Secondary Outcome: Cumulative Probability of Infant HIV-infection
Description: The Kaplan-Meier estimate of the cumulative probability of infants acquiring HIV-1 infection from birth through 50 weeks after birth based on nucleic acid test results.
Time Frame: Birth through 50 weeks after birth
Population: Live born infants
Measure: Number; unit: Cumulative probability per 100 persons
Arm/Group | Arm 1 Infants | Arm 2 Infants | Arm 3 Infants
Number analyzed (Participants) | 208 | 202 | 207
Cumulative probability per 100 persons | 0.98 | 0.50 | 0.55
Statistical Analysis 1: Comparison: Arm 1 Infants vs Arm 2 Infants; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.28, Z-test; Risk Difference (RD) = 0.5, 95% CI 2-sided [-1.2 to 2.1]
Statistical Analysis 2: Comparison: Arm 2 Infants vs Arm 3 Infants; The Kaplan-Meier method was used to estimate survival probabilities. Survival probabilities were compared based on a Z-test using Greenwoods estimate of the standard error. The null hypothesis was no difference between arms (DTG+FTC/TDF - EFV/FTC/TDF); Test type: Superiority; p = 0.47, Z-test; Risk Difference (RD) = -0.1, 95% CI 2-sided [-1.5 to 1.4]
Statistical Analysis 3: Comparison: Arm 1 Infants vs Arm 3 Infants; The Kaplan-Meier method was used to estimate survival probabilities. Survival probabilities were compared based on a Z-test using Greenwoods estimate of the standard error. The null hypothesis was no difference between arms (DTG+FTC/TAF - EFV/FTC/TDF); Test type: Superiority; p = 0.31, Z-test; Risk Difference (RD) = 0.4, 95% CI 2-sided [-1.3 to 2.2]

16. Secondary Outcome: Cumulative Probability of Infant Deaths
Description: The Kaplan-Meier estimate of the cumulative probability of infant deaths from birth through 50 weeks after birth.
Time Frame: Birth through 50 weeks after birth
Population: Live born infants
Measure: Number; unit: Cumulative probability per 100 persons
Arm/Group | Arm 1 Infants | Arm 2 Infants | Arm 3 Infants
Number analyzed (Participants) | 208 | 202 | 207
Cumulative probability per 100 persons | 1.0 | 2.0 | 6.9
Statistical Analysis 1: Comparison: Arm 1 Infants vs Arm 2 Infants; Test type: Superiority — The Kaplan-Meier method was used to estimate survival probabilities. Comparisons of survival probabilities was based on a Z-test using Greenwoods estimate of the standard error. The null hypothesis was no difference between arms, with estimated difference of DTG+FTC/TAF - DTG+FTC/TDF; p = 0.20, Z-test; Risk Difference (RD) = -1.0, 95% CI 2-sided [-3.4 to 1.3]
Statistical Analysis 2: Comparison: Arm 2 Infants vs Arm 3 Infants; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.008, Z-test; Risk Difference (RD) = -4.9, 95% CI 2-sided [-8.9 to -0.9]
Statistical Analysis 3: Comparison: Arm 1 Infants vs Arm 3 Infants; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p < 0.001, Z-test; Risk Difference (RD) = -5.9, 95% CI 2-sided [-9.7 to -2.2]

17. Secondary Outcome: Maternal Change in Creatinine Clearance
Description: Maternal change in creatinine clearance per week based on generalized estimating equations
Time Frame: Baseline to 50 weeks postpartum
Population: Women with creatinine clearance data.
Measure: Mean (95% Confidence Interval); unit: mL/min
Arm/Group | Arm 1: Maternal DTG+FTC/TAF | Arm 2: Maternal DTG+FTC/TDF | Arm 3: Maternal EFV/FTC/TDF
Number analyzed (Participants) | 215 | 214 | 210
mL/min | -0.980 [-1.066 to -0.894] | -0.887 [-0.964 to -0.810] | -0.935 [-1.013 to -0.857]
Statistical Analysis 1: Comparison: Arm 1: Maternal DTG+FTC/TAF vs Arm 2: Maternal DTG+FTC/TDF; Null hypothesis of no difference in weekly change in creatinine clearance from baseline (DTG+FTC/TAF - DTG+FTC/TDF); Test type: Superiority; p = 0.12, Generalized Estimating Equation; Mean Difference (Final Values) = -0.093, 95% CI 2-sided [-0.208 to 0.023]
Statistical Analysis 2: Comparison: Arm 2: Maternal DTG+FTC/TDF vs Arm 3: Maternal EFV/FTC/TDF; Null hypothesis of no difference in weekly change in creatinine clearance from baseline (DTG+FTC/TDF - EFV/FTC/TDF); Test type: Superiority; p = 0.39, Generalized Estimating Equation; Mean Difference (Final Values) = 0.048, 95% CI 2-sided [-0.061 to 0.158]
Statistical Analysis 3: Comparison: Arm 1: Maternal DTG+FTC/TAF vs Arm 3: Maternal EFV/FTC/TDF; Null hypothesis of no difference in weekly change in creatinine clearance from baseline (DTG+FTC/TAF - EFV/FTC/TDF); Test type: Superiority; p = 0.45, Generalized Estimating Equation; Mean Difference (Final Values) = -0.045, 95% CI 2-sided [-0.161 to 0.072]

18. Secondary Outcome: Infant Creatinine Clearance
Description: Infant creatinine clearance based on Schwartz formula
Time Frame: Delivery and 26 weeks postpartum
Population: Live born infants with creatinine clearance data
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Arm 1 Infants | Arm 2 Infants | Arm 3 Infants
Number analyzed (Participants) | 193 | 189 | 185
mL/min
  Delivery | 52.7 (29.6) | 53.1 (69.7) | 49.0 (24.7)
  26 Weeks Postpartum | 134.8 (109.6) | 123.6 (40.3) | 135.0 (51.1)
Statistical Analysis 1: Comparison: Arm 1 Infants vs Arm 2 Infants; Null hypothesis of no difference between arms at delivery (DTG+FTC/TAF - DTG+FTC/TDF); Test type: Superiority; p = 0.94, t-test, 2 sided; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-11.3 to 10.5]
Statistical Analysis 2: Comparison: Arm 2 Infants vs Arm 3 Infants; Null hypothesis of no difference between arms at delivery (DTG+FTC/TDF - EFV/FTC/TDF); Test type: Superiority; p = 0.44, t-test, 2 sided; Mean Difference (Final Values) = 4.2, 95% CI 2-sided [-6.5 to 14.9]
Statistical Analysis 3: Comparison: Arm 1 Infants vs Arm 3 Infants; Null hypothesis of no difference between arms at delivery (DTG+FTC/TAF - EFV/FTC/TDF); Test type: Superiority; p = 0.18, t-test, 2 sided; Mean Difference (Final Values) = 3.8, 95% CI 2-sided [-1.8 to 9.3]
Statistical Analysis 4: Comparison: Arm 1 Infants vs Arm 2 Infants; Null hypothesis of no difference between arms at week 26 (DTG+FTC/TAF - DTG+FTC/TDF); Test type: Superiority; p = 0.27, t-test, 2 sided; Mean Difference (Final Values) = 11.1, 95% CI 2-sided [-8.9 to 31.1]
Statistical Analysis 5: Comparison: Arm 2 Infants vs Arm 3 Infants; Null hypothesis of no difference between arms at week 26 (DTG+FTC/TDF - EFV/FTC/TDF); Test type: Superiority; p = 0.048, t-test, 2 sided; Mean Difference (Final Values) = -11.4, 95% CI 2-sided [-22.6 to -0.1]
Statistical Analysis 6: Comparison: Arm 1 Infants vs Arm 3 Infants; Null hypothesis of no difference between arms at week 26 (DTG+FTC/TAF - EFV/FTC/TDF); Test type: Superiority; p = 0.98, t-test, 2 sided; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-21.0 to 20.5]

19. Secondary Outcome: Percentage of Mothers With HIV-1 ARV Drug Resistance Mutations at the Time of Maternal Virologic Failure
Description: Percentage of mothers with HIV-1 antiretroviral (ARV) drug resistance mutations at the time of maternal virologic failure. Virologic failure was defined as two consecutive plasma HIV-1 RNA viral loads <200 copies/mL on or after 24 weeks on study. Drug resistance mutations were assessed using the Stanford algorithm, and all ARV regimens were assessed for mutations.
Time Frame: From 24 weeks after randomization through Week 50 postpartum
Population: All enrolled women
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Maternal DTG+FTC/TAF | Arm 2: Maternal DTG+FTC/TDF | Arm 3: Maternal EFV/FTC/TDF
Number analyzed (Participants) | 217 | 215 | 211
percentage of participants | 0.92 | 1.86 | 6.16
Statistical Analysis 1: Comparison: Arm 1: Maternal DTG+FTC/TAF vs Arm 2: Maternal DTG+FTC/TDF; Null hypothesis of no difference between groups (DTG+FTC/TAF - DTG+FTC/TDF); Test type: Superiority; p = 0.40, Wald test of two proportions; Risk Difference (RD) = -0.9, 95% CI 2-sided [-3.1 to 1.3]
Statistical Analysis 2: Comparison: Arm 2: Maternal DTG+FTC/TDF vs Arm 3: Maternal EFV/FTC/TDF; Null hypothesis of no difference between groups (DTG+FTC/TDF - EFV/FTC/TDF); Test type: Superiority; p = 0.023, Wald test of two proportions; Risk Difference (RD) = -4.3, 95% CI 2-sided [-8.0 to -0.6]
Statistical Analysis 3: Comparison: Arm 1: Maternal DTG+FTC/TAF vs Arm 3: Maternal EFV/FTC/TDF; Null hypothesis of no difference between groups (DTG+FTC/TAF - EFV/FTC/TDF); Test type: Superiority; p = 0.003, Wald test of two proportions; Risk Difference (RD) = -5.2, 95% CI 2-sided [-8.7 to -1.8]

20. Secondary Outcome: Count of Infants With HIV-1 Antiretroviral Drug Resistance Mutations at the Time of Infant HIV Diagnosis
Description: Count of infants with HIV-1 antiretroviral drug resistance mutations (to any antiretroviral drug) at the time of infant HIV diagnosis, based on laboratory blood test results.
Time Frame: From birth through 50 weeks postpartum
Population: Infants who had an HIV diagnosis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Infants | Arm 2 Infants | Arm 3 Infants
Number analyzed (Participants) | 2 | 1 | 1
Participants | 1 | 0 | 1

21. Secondary Outcome: Percentage of Mother-Infant Pairs With Preterm Deliveries
Description: Percentage of mother-infant pairs with preterm deliveries (<37 weeks gestation) resulting in live born infant
Time Frame: Delivery
Population: Women with pregnancies resulting in a live born infant
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Maternal DTG+FTC/TAF | Arm 2: Maternal DTG+FTC/TDF | Arm 3: Maternal EFV/FTC/TDF
Number analyzed (Participants) | 208 | 202 | 207
percentage of participants | 5.8 | 9.4 | 12.1
Statistical Analysis 1: Comparison: Arm 1: Maternal DTG+FTC/TAF vs Arm 2: Maternal DTG+FTC/TDF; Test type: Non-Inferiority — Equivalence margin was a 10% difference between groups; p = 0.16, Wald test of two proportions; Risk Difference (RD) = -3.6, 95% CI 2-sided [-8.8 to 1.5]
Statistical Analysis 2: Comparison: Arm 2: Maternal DTG+FTC/TDF vs Arm 3: Maternal EFV/FTC/TDF; Test type: Non-Inferiority — Equivalence margin was a 10% difference between groups; p = 0.38, Wald test of two proportions; Risk Difference (RD) = -2.7, 95% CI 2-sided [-8.7 to 3.3]
Statistical Analysis 3: Comparison: Arm 1: Maternal DTG+FTC/TAF vs Arm 3: Maternal EFV/FTC/TDF; Test type: Non-Inferiority — Equivalence margin was a 10% difference between groups; p = 0.023, Wald test of two proportions; Risk Difference (RD) = -6.3, 95% CI 2-sided [-11.8 to -0.9]

22. Secondary Outcome: Percentage of Infants Born Small for Gestational Age
Description: Percentage of infants born small for gestational age (<10th percentile adjusted for sex assigned at birth) based on Intergrowth 21st Standards
Time Frame: Birth
Population: Live born infants with weight and sex data available.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 Infants | Arm 2 Infants | Arm 3 Infants
Number analyzed (Participants) | 202 | 200 | 200
percentage of participants | 16.3 | 22.5 | 20.5
Statistical Analysis 1: Comparison: Arm 1 Infants vs Arm 2 Infants; Test type: Non-Inferiority — Equivalence margin was a 10% difference between groups; p = 0.12, Wald test of two proportions; Risk Difference (RD) = -6.2, 95% CI 2-sided [-13.9 to 1.5]
Statistical Analysis 2: Comparison: Arm 2 Infants vs Arm 3 Infants; Test type: Non-Inferiority — Equivalence margin was a 10% difference between groups; p = 0.63, Wald test of two proportions; Risk Difference (RD) = 2.0, 95% CI 2-sided [-6.0 to 10.0]
Statistical Analysis 3: Comparison: Arm 1 Infants vs Arm 3 Infants; Test type: Non-Inferiority — Equivalence margin was a 10% difference between groups; p = 0.28, Wald test of two proportions; Risk Difference (RD) = -4.2, 95% CI 2-sided [-11.7 to 3.4]

23. Secondary Outcome: Change in Maternal Weight Antepartum
Description: Change in maternal antepartum weight per week based on generalized estimating equations
Time Frame: Baseline through before delivery (up to one day prior)
Population: Women with weight data available.
Measure: Mean (95% Confidence Interval); unit: kg/week
Arm/Group | Arm 1: Maternal DTG+FTC/TAF | Arm 2: Maternal DTG+FTC/TDF | Arm 3: Maternal EFV/FTC/TDF
Number analyzed (Participants) | 217 | 215 | 210
kg/week | 0.378 [0.343 to 0.412] | 0.319 [0.291 to 0.348] | 0.291 [0.260 to 0.322]
Statistical Analysis 1: Comparison: Arm 1: Maternal DTG+FTC/TAF vs Arm 2: Maternal DTG+FTC/TDF; Null hypothesis of no difference between arms (DTG+FTC/TAF - DTG+FTC/TDF); Test type: Superiority; p = 0.011, Generalized Estimating Equation; Mean Difference (Final Values) = 0.058, 95% CI 2-sided [0.013 to 0.103]
Statistical Analysis 2: Comparison: Arm 2: Maternal DTG+FTC/TDF vs Arm 3: Maternal EFV/FTC/TDF; Null hypothesis of no difference between arms (DTG+FTC/TDF - EFV/FTC/TDF); Test type: Superiority; p = 0.19, Generalized Estimating Equation; Mean Difference (Final Values) = 0.028, 95% CI 2-sided [-0.014 to 0.070]
Statistical Analysis 3: Comparison: Arm 1: Maternal DTG+FTC/TAF vs Arm 3: Maternal EFV/FTC/TDF; Null hypothesis of no difference between arms (DTG+FTC/TAF - EFV/FTC/TDF); Test type: Superiority; p < 0.001, Generalized Estimating Equation; Mean Difference (Final Values) = 0.086, 95% CI 2-sided [0.040 to 0.133]

24. Secondary Outcome: Change in Maternal Weight Postpartum
Description: Change in maternal postpartum weight per week based on generalized estimating equations
Time Frame: Delivery to 50 weeks postpartum
Population: Women with weight data available.
Measure: Mean (95% Confidence Interval); unit: kg/week
Arm/Group | Arm 1: Maternal DTG+FTC/TAF | Arm 2: Maternal DTG+FTC/TDF | Arm 3: Maternal EFV/FTC/TDF
Number analyzed (Participants) | 212 | 212 | 207
kg/week | 0.014 [-0.004 to 0.032] | -0.008 [-0.027 to 0.012] | -0.032 [-0.048 to -0.017]
Statistical Analysis 1: Comparison: Arm 1: Maternal DTG+FTC/TAF vs Arm 2: Maternal DTG+FTC/TDF; Null hypothesis of no difference between arms (DTG+FTC/TAF - DTG+FTC/TDF); Test type: Superiority; p = 0.11, Generalized Estimating Equation; Mean Difference (Final Values) = 0.022, 95% CI 2-sided [-0.005 to 0.048]
Statistical Analysis 2: Comparison: Arm 2: Maternal DTG+FTC/TDF vs Arm 3: Maternal EFV/FTC/TDF; Null hypothesis of no difference between arms (DTG+FTC/TDF - EFV/FTC/TDF); Test type: Superiority; p = 0.055, Generalized Estimating Equation; Mean Difference (Final Values) = 0.024, 95% CI 2-sided [-0.000 to 0.049]
Statistical Analysis 3: Comparison: Arm 1: Maternal DTG+FTC/TAF vs Arm 3: Maternal EFV/FTC/TDF; Null hypothesis of no difference between arms (DTG+FTC/TAF - EFV/FTC/TDF); Test type: Superiority; p < 0.001, Generalized Estimating Equation; Mean Difference (Final Values) = 0.046, 95% CI 2-sided [0.022 to 0.070]

25. Secondary Outcome: Change in Maternal Weight Overall
Description: Change in maternal weight per week based on generalized estimating equations
Time Frame: Baseline to 50 weeks postpartum
Population: Women with weight data available.
Measure: Mean (95% Confidence Interval); unit: kg/week
Arm/Group | Arm 1: Maternal DTG+FTC/TAF | Arm 2: Maternal DTG+FTC/TDF | Arm 3: Maternal EFV/FTC/TDF
Number analyzed (Participants) | 217 | 215 | 211
kg/week | -0.027 [-0.042 to -0.012] | -0.050 [-0.066 to -0.034] | -0.084 [-0.098 to -0.070]
Statistical Analysis 1: Comparison: Arm 1: Maternal DTG+FTC/TAF vs Arm 2: Maternal DTG+FTC/TDF; Null hypothesis of no difference between arms (DTG+FTC/TAF - DTG+FTC/TDF); Test type: Superiority; p = 0.041, Generalized Estimating Equation; Mean Difference (Final Values) = 0.023, 95% CI 2-sided [0.001 to 0.045]
Statistical Analysis 2: Comparison: Arm 2: Maternal DTG+FTC/TDF vs Arm 3: Maternal EFV/FTC/TDF; Null hypothesis of no difference between arms (DTG+FTC/TDF - EFV/FTC/TDF); Test type: Superiority; p = 0.002, Generalized Estimating Equation; Mean Difference (Final Values) = 0.034, 95% CI 2-sided [0.013 to 0.055]
Statistical Analysis 3: Comparison: Arm 1: Maternal DTG+FTC/TAF vs Arm 3: Maternal EFV/FTC/TDF; Null hypothesis of no difference between arms (DTG+FTC/TAF - EFV/FTC/TDF); Test type: Superiority; p < 0.001, Generalized Estimating Equation; Mean Difference (Final Values) = 0.057, 95% CI 2-sided [0.036 to 0.078]

ADVERSE EVENTS:
Time Frame: For women, adverse events were reported from randomization through study visit occurring at 50 weeks postpartum. For infants, adverse events were reported from birth through the study visit occurring at 50 weeks post birth.
Description: All grade 3 or higher and serious adverse events were reported. Other targeted lower grade adverse events. All randomized women and live born infants were summarized. The DAIDS AE Grading Table, Corrected Version 2.1, dated July 2017, was used in this study. A full description of adverse event data collection is provided in protocol Section 7.2.
Arm/Group | Arm 1: Maternal DTG+FTC/TAF | Arm 2: Maternal DTG+FTC/TDF | Arm 3: Maternal EFV/FTC/TDF | Arm 1 Infants | Arm 2 Infants | Arm 3 Infants
All-Cause Mortality (participants affected / at risk) | 1/217 | 0/215 | 0/211 | 2/208 | 4/202 | 14/207
Serious Adverse Events (participants affected / at risk) | 39/217 | 39/215 | 40/211 | 35/208 | 29/202 | 44/207
Other Adverse Events (participants affected / at risk) | 189/217 | 198/215 | 143/211 | 34/208 | 40/202 | 34/207
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Maternal DTG+FTC/TAF (N=217) | Arm 2: Maternal DTG+FTC/TDF (N=215) | Arm 3: Maternal EFV/FTC/TDF (N=211) | Arm 1 Infants (N=208) | Arm 2 Infants (N=202) | Arm 3 Infants (N=207)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1 | 0 | 0
Anaemia neonatal (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anaemia of pregnancy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia neonatal (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia neonatal (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Accessory auricle (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anomalous pulmonary venous connection (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arachnodactyly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 3 | 0 | 0
Congenital foot malformation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0
Congenital inguinal hernia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1
Congenital joint malformation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1
Congenital mitral valve incompetence (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0
Congenital skin dimples (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 2 | 0 | 0
Congenital syphilis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 1 | 1
Congenital tricuspid valve incompetence (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0
Congenital ureteric anomaly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0
Duodenal atresia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haemangioma congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1
Macrocephaly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0
Multiple congenital abnormalities (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0
Naevus flammeus (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sickle cell anaemia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sickle cell disease (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0
Talipes (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 1
Ileal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Infantile vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Death neonatal (General disorders) | 0 | 0 | 0 | 0 | 1 | 3
Fever neonatal (General disorders) | 0 | 0 | 0 | 2 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Amniotic cavity infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 3
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Disseminated tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 2
Malaria (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Meningitis pneumococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Neonatal pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1
Pelvic inflammatory disease (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 4 | 2 | 5
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1
Postoperative wound infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Postpartum sepsis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pyometra (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Sepsis neonatal (Infections and infestations) | 0 | 0 | 0 | 4 | 7 | 6
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Staphylococcal scalded skin syndrome (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2
Tracheobronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 3 | 2 | 0 | 1 | 1
Urinary tract infection neonatal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Wound sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Uterine rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac murmur (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 3 | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypoglycaemia neonatal (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Fontanelle bulging (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 5
Infant irritability (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Intraventricular haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neonatal seizure (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 | 1 | 2 | 0 | 0 | 0
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0
Birth trauma (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1
Cervix dystocia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 | 0 | 0 | 0
Failed induction of labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0
Failed trial of labour (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0
False labour (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0 | 0 | 0 | 0
Foetal death (Pregnancy, puerperium and perinatal conditions) | 6 | 7 | 1 | 0 | 0 | 0
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 2 | 2 | 5 | 0 | 0 | 0
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0 | 0 | 0 | 0
Foetal hypokinesia (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 4 | 5 | 7 | 0 | 0 | 0
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 1 | 2 | 0 | 0 | 0
Hydrops foetalis (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0
Hypothermia neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0
Imminent abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 1 | 0
Large for dates baby (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 1 | 0
Meconium in amniotic fluid (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 1
Neonatal disorder (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 0
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 0 | 3 | 1 | 0 | 0 | 0
Placenta praevia (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 3 | 0 | 0 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 4 | 2 | 0 | 0 | 0 | 0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 5 | 4
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 4 | 1 | 1 | 0 | 0 | 0
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 3 | 1 | 1 | 0 | 0 | 0
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0 | 0 | 0 | 0
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 2 | 3 | 4 | 0 | 0 | 0
Prolonged labour (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1 | 0 | 0 | 0
Prolonged pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0
Prolonged rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0 | 0 | 0 | 0
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 1 | 2 | 3 | 0 | 0 | 0
Threatened labour (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 0 | 0 | 0 | 0
Umbilical cord around neck (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0
Umbilical cord cyst (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0
Umbilical cord prolapse (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 | 0 | 0 | 0
Uterine atony (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0
Alcoholism (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pyelocaliectasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Grunting (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Meconium aspiration syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 5
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 1 | 2
Neonatal respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 5 | 2 | 2
Neonatal tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 0 | 1
Use of accessory respiratory muscles (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash neonatal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Physical assault (Social circumstances) | 0 | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Essential hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Maternal DTG+FTC/TAF (N=217) | Arm 2: Maternal DTG+FTC/TDF (N=215) | Arm 3: Maternal EFV/FTC/TDF (N=211) | Arm 1 Infants (N=208) | Arm 2 Infants (N=202) | Arm 3 Infants (N=207)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 3 | 0 | 0 | 1
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anaemia of pregnancy (Blood and lymphatic system disorders) | 3 | 2 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 2 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Congenital joint malformation (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0
Congenital toxoplasmosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0
Congenital umbilical hernia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 1
Polydactyly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 2
Trisomy 21 (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Developmental delay (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Macrosomia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 2 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Immune reconstitution inflammatory syndrome (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Amniotic cavity infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Furuncle (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Genital herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Impetigo (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Perihepatitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Postpartum sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Sepsis neonatal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Skin bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Tracheobronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Tuberculous pleurisy (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Vulvovaginitis trichomonal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 5 | 6 | 4 | 0 | 0 | 0
Amylase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 4 | 4 | 0 | 0 | 0
Bilirubin conjugated increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 170 | 179 | 76 | 4 | 8 | 4
Blood glucose decreased (Investigations) | 0 | 0 | 0 | 3 | 2 | 4
Blood pressure increased (Investigations) | 2 | 1 | 1 | 0 | 0 | 0
Blood sodium decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Creatinine renal clearance decreased (Investigations) | 182 | 193 | 132 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 8 | 20 | 14 | 8 | 8 | 7
Head lag (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 2 | 10 | 7 | 14
Neutrophil count increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 1 | 0 | 3 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Poor feeding infant (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Underweight (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Neonatal seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Poor sucking reflex (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 2 | 2 | 0 | 0 | 0 | 0
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 3 | 0 | 0 | 0
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 2 | 1 | 1
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 2 | 1 | 1
Meconium in amniotic fluid (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0
Morning sickness (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 2 | 0 | 0 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 2 | 2 | 0 | 0 | 0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1 | 1
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 1 | 0 | 0 | 0
Premature labour (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0
Prolonged pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 3 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Perinatal depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neonatal asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neonatal respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neonatal tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Transient tachypnoea of the newborn (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urticaria papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abortion induced (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0
Caesarean section (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 1 | 2 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights

DOCUMENTS (5):
  • Study Protocol and Informed Consent Form: IMPAACT 2010 Protocol V2.0 (2017-12-08): https://cdn.clinicaltrials.gov/large-docs/22/NCT03048422/Prot_ICF_000.pdf
  • Study Protocol: IMPAACT 2010 Protocol V2.0_Letter of Amendment 1 (2018-07-20): https://cdn.clinicaltrials.gov/large-docs/22/NCT03048422/Prot_001.pdf
  • Study Protocol: IMPAACT 2010 Protocol V2.0_Letter of Amendment 2 (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/22/NCT03048422/Prot_002.pdf
  • Study Protocol: IMPAACT 2010 Protocol V2.0_Letter of Amendment 3 (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/22/NCT03048422/Prot_003.pdf
  • Statistical Analysis Plan (2020-10-26): https://cdn.clinicaltrials.gov/large-docs/22/NCT03048422/SAP_004.pdf